CLINICAL TRIAL: NCT06923722
Title: A Placebo-controlled, Randomized, Double-masked, Cross-over Acute Intervention Study Investigating the Effects of Grape Polyphenols on Cerebral Oxygenation, Cognitive and Vascular Function in the Context of Mental Stress in Young Adults
Brief Title: De-stressing the Brain: Can Eating Grapes During Periods of Mental Stress Protect Brain and Vascular Health in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Catarina Rendeiro, Principal Investigator, Assistant Professor in Nutritional Sciences, University of Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ERN_17-1755H; 3155902 (Other Grant/Funding Number: California Table Grape Comission)
Record Dates: First submitted 2025-03-27; First posted 2025-04-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: vascular function; flavonoids; cerebral oxygenation; mental stress; cognition; executive function; grape; Flow-mediated dilatation; Functional Near-Infrared Spectroscopy
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The interventions have been masked by the intervention supplier (California Table Grape Commission). Therefore, all researchers are blinded to the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flavonoid grape intervention (Experimental): 60 g freeze-dried grape powder, equivalent to 300 g fresh grapes (Total polyphenols: 437 mg/100g)
  Interventions: Dietary Supplement: High-flavonoid grape intervention
- Low-flavonoid grape intervention (Placebo Comparator): 60 g powder isocaloric-matched control (Total polyphenols: < 60 mg)
  Interventions: Dietary Supplement: Low-flavonoid grape intervention

INTERVENTIONS:
Dietary Supplement: High-flavonoid grape intervention — High-flavonoid grape powder: 60 g, equivalent to 300 g fresh grapes. Total polyphenols: 437 mg/100g).
  Arms: High-flavonoid grape intervention
Dietary Supplement: Low-flavonoid grape intervention — 60 g powder isocaloric-matched control (Total polyphenols: < 60 mg)
  Arms: Low-flavonoid grape intervention

SUMMARY:
The main aim of the current study is to investigate whether consuming grapes rich in flavonoids just before mental stress can protect cerebrovascular and peripheral vascular function, mood and cognition, from the negative effects of mental stress in young healthy adults. A second, exploratory aim, will further address whether quality of habitual diet, microbiome health (composition; metabolites production e.g. Short-chain fatty acids) and levels of cardiorespiratory fitness play a role on the beneficial effects of grapes during mental stress. All participants will receive a high-flavonoid grape intervention (60 g freeze-dried grape powder, equivalent to 300 g fresh grapes) and a low-flavonoid grape intervention (60 g powdere isocaloric-matched control). It is hypothesized that the high-flavonoid grape intervention will improve cortical oxygenation and cognitive function in the context of mental stress, and prevent the stress-induced decline in peripheral endothelial function following stress. Furthermore, it is hypothesized that individuals with poorer diets, cardiorespiratory fitness and a poorer gut microbiome will benefit more from the grape intervention in the context of mental stress.

DETAILED DESCRIPTION:
Psychological stress is widespread in our societies, and has been extensively shown to have negative consequences for human health. Specifically, psychological stress induces significant declines in human vascular function, as measured by brachial Flow-mediated Dilatation (FMD). We have demonstrated that flavonoid interventions can prevent the harmful effects of stress on the vascular system. Indeed, flavonoid-rich interventions have also been extensively shown to improve peripheral and cerebrovascular function in the absence of stress. However, the effect of flavonoids on cerebrovascular function and cognition in the context of mental stress is unknown. In the proposed project, our key objectives are to investigate whether grape intake prior to a mental stress task results in better brain oxygenation and vascular function, which leads to improved cognitive performance and mood in young healthy adults. These data will establish whether grapes can be effective as a 'stress snack' to optimize cognitive and brain function in the context of psychological stress. Furthermore, we will explore whether there are certain participant characteristics that mediate the impact of grape flavonoids on cerebrovascular function and cognition in the context of mental stress. Such as, physical fitness (assessed by a VO2 max test), composition of gut microbiome (assessed by faecal sample), habitual diet (assessed by 3-day food diary and the food frequency questionnaire), and eating behaviour and chronic stress (assessed by the eating behaviour questionnaire and perceived stress scale). This work will be important to guide future dietary recommendations around stress and might ultimately result in increased intake of flavonoid-rich grapes and other flavonoid-rich fruits/vegetables overall.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 - 40 years old

Exclusion Criteria:

* Smokers
* Consumes > 21 units of alcohol per week
* History of cardiovascular, respiratory, metabolic, liver or inflammatory diseases
* Suffers from blood-clotting disorders
* Allergies or intolerances to foods
* On a weight reducing dietary regiment
* Currently taking dietary supplements, including fatty acids and vitamins
* On long-term medication or have been on antibiotics in the last 3 months
* Has an infection at present (e.g. cold) or viral infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pre-frontal cortical Tissue Oxygenation Index (NIRS) - TOI | Change from pre-intervention baseline to 1 hour post-intervention (during mental stress) and 1 hour 15 minutes post-intervention (during cognitive tasks, 10 minutes post-stress)
  Pre-frontal levels of Tissue Oxygenation Index (% TOI) will be assessed by functional Near-Infrared Spectroscopy (fNIRS). The NIRS device measures changes in chromophore concentrations of oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb), providing depth-resolved measures of total tissue oxygen saturation.
Pre-frontal cortical Tissue Oxygenation Index (NIRS) - O2Hb | Change from pre-intervention baseline to 1 hour post-intervention (during mental stress) and 1 hour 15 minutes post-intervention (during cognitive tasks, 10 minutes post-stress).
  Pre-frontal levels of oxygenated (O2Hb) haemoglobin concentration (μmol) will be assessed by functional Near-Infrared Spectroscopy (fNIRS).
Pre-frontal cortical Tissue Oxygenation Index (NIRS) - HHb | Change from pre-intervention baseline to 1 hour post-intervention (during mental stress) and 1 hour 15 minutes post-intervention (during cognitive tasks, 10 minutes post-stress).
  Pre-frontal levels of deoxygenated (HHb) haemoglobin concentration (μmol) will be assessed by functional Near-Infrared Spectroscopy (fNIRS).
Pre-frontal cortical Tissue Oxygenation Index (NIRS) - nTHI | Change from pre-intervention baseline to 1 hour post-intervention (during mental stress) and 1 hour 15 minutes post-intervention (during cognitive tasks, 10 minutes post-stress).
  Pre-frontal levels of normalised haemoglobin index (relative value of total haemoglobin normalised to the initial value, nTHI) content (a.u.) will be assessed by functional Near-Infrared Spectroscopy (fNIRS).

SECONDARY OUTCOMES:
Flow-mediated dilatation (FMD) of the brachial artery | Change from pre-intervention baseline to 2 hours and 2 hours 45 minutes post-intervention (45-90 minutes post-stress).
  FMD of the brachial artery. Expressed as % FMD: change in brachial diameter from baseline to peak dilation following 5 minutes of arterial occlusion. Brachial artery diameter and blood flow will be measured using Doppler ultrasonography (uSmart 3300, Terason).
Common Carotid Artery (CCA) - Blood flow | Change from pre-intervention baseline to 2 hours and 2 hours 45 minutes post-intervention (45-90 minutes post-stress).
  Common Carotid Artery (CCA) blood flow velocity (ml min-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software. CCA blood flow is calculated using CCA blood velocity and diameter across 2 minutes of recording.
Common Carotid Artery (CCA) - Shear rate | Change from pre-intervention baseline to 2 hours and 2 hours 45 minutes post-intervention (45-90 minutes post-stress).
  Common Carotid Artery (CCA) shear rate (s-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software.
Executive Function (MANT) - Accuracy | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function accuracy will be measured using the Modified Attention Network Task (MANT) which measures response to cognitive load
Executive Function (Switch) - Accuracy | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function accuracy will be measured using the Switch Task which considers cognitive flexibility.
Executive Function (MANT) - Reaction time | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function reaction time will be measured using Modified Attention Network Task (MANT) which measures response to cognitive load.
Executive Function (Switch) - Reaction time | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function reaction time will be measured using the Switch Task which considers cognitive flexibility.
Executive Function (MANT) - Inverse Efficiency Score | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function inverse efficiency will be measured using the Modified Attention Network Task (MANT), calculated by dividing task reaction time by task accuracy.
Executive Function (Switch) - Inverse Efficiency Score | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress).
  Executive function inverse efficiency will be measured using the Switch Task, calculated by dividing task reaction time by task accuracy.
Mood (POMS) | Change from pre-intervention baseline to 1 hour post-intervention (immediately following stress), 2 hours and 2 hours 45 minutes post-intervention (45-90 minutes post-stress).
  Mood (total mood disturbance, TMD) will be assessed by the questionnaire Profile-of-Mood-States (POMS).

OTHER OUTCOMES:
Forearm blood flow (FBF) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Venous occlusion plethysmography will assess the forearm vasodilatory response (ml/100ml/min) to mental stress.
Forearm vascular conductance (FVC) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Forearm vascular conductance (FVC) will be calculated by dividing FBF by beat-to-beat mean arterial pressure (MAP).
Cardiovascular activity - Heart rate (HR) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Heart rate (HR, bpm) is assessed using an electrocardiogram.
Cardiovascular activity - R-wave to pulse interval (RPI) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  R-wave to pulse interval (RPI, ms) is assessed using an electrocardiogram, to provide an indication of sympathetic activity.
Cardiovascular activity - Heart rate variability (HRV) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Heart rate variability (HRV, ms) is assessed using an electrocardiogram, to provide an indication of parasympathetic activity.
Cardiovascular activity - beat-to-beat systolic blood pressure (SBP) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Beat-to-beat systolic blood pressure (SBP) will be measured using a Finometer (mmHg).
Cardiovascular activity - beat-to-beat diastolic blood pressure (DBP) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Beat-to-beat diastolic blood pressure (SBP) will be measured using a Finometer (mmHg).
Cardiovascular activity - beat-to-beat mean arterial pressure (MAP) | Change from pre-intervention baseline to 1 hour post-intervention (during 8 minutes rest and 8 minutes of mental stress).
  Beat-to-beat mean arterial pressure (MAP) will be measured using a Finometer (mmHg).
Brachial Systolic Blood Pressure (SBP) | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress), 2 hours post-intervention (45 minutes post-stress) and 2 hour 45 minutes post-intervention (90 minutes post-stress).
  Resting systolic blood pressure (mmHg) will be measured using an automated oscillometric blood pressure monitor, with a cuff attached to the right upper arm, following at least 10 minutes rest.
Brachial Diastolic Blood Pressure (DBP) | Change from pre-intervention baseline to 1 hour 15 minutes post-intervention (10 minutes post-stress), 2 hours post-intervention (45 minutes post-stress) and 2 hour 45 minutes post-intervention (90 minutes post-stress).
  Resting diastolic blood pressure (mmHg) will be measured using an automated oscillometric blood pressure monitor, with a cuff attached to the right upper arm, following at least 10 minutes rest.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise & Rehabilitation Sciences, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No